CLINICAL TRIAL: NCT04652362
Title: A Single-session Growth Mindset Intervention for Children and Young People With Mental Health Difficulties: a Randomised Controlled Trial
Brief Title: A Single-session Growth Mindset Intervention for Children and Young People With Mental Health Difficulties
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Lead researcher off sick
Sponsor: Royal Holloway University (Other)
Responsible Party: Principal Investigator, Harriet Clarkson, Trainee Clinical Psychologist, Royal Holloway University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2243
Record Dates: First submitted 2020-11-26; First posted 2020-12-03 (Actual); Last update posted 2022-05-12 (Actual); Status verified 2022-05

CONDITIONS: Anxiety; Anxiety Disorders; Depression; Low Mood
Keywords: controlled clinical trials; internet-based intervention
MeSH Terms: conditions — Anxiety Disorders; Depression; Consciousness Disorders

STUDY DESIGN:
Intervention Model Description: Participants will be randomly allocated to either the growth mindset intervention or the supportive therapy control condition.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participants will not be informed about the contents of the two different programmes and therefore will be blind to group allocation. Randomisation, questionnaire and intervention delivery will be fully automated through the Qualtrics platform and therefore researchers will also be blind to group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Growth Mindset Intervention (Experimental)
  Interventions: Behavioral: Growth Mindset Online Single-Session Intervention
- Supportive Therapy Intervention (Active Comparator)
  Interventions: Behavioral: Supportive Therapy Online Single-Session Intervention (Control)

INTERVENTIONS:
Behavioral: Growth Mindset Online Single-Session Intervention — During the self-administered single session intervention participants are provided with basic information about the brain and are introduced to the concept of neuroplasticity. The concept of neuroplasticity is applied to personal traits, such as shyness, anxiety and sadness, and young people are taught that these traits are the result of thoughts and feelings in our brain and are amenable to change. Participants are presented with scientific information and research evidence to support the idea that people have the potential to change and are given vignettes from older children detailing how they have used a growth mindset to overcome difficulties. The intervention takes approximately 20-30 minutes to complete.
  Arms: Growth Mindset Intervention
Behavioral: Supportive Therapy Online Single-Session Intervention (Control) — The single session supportive therapy intervention was designed to be structurally comparable to the growth mindset intervention, including the same number of reading and writing activities. Participants were provided with information about emotions and the benefits of expressing emotions. Vignettes from older children described times they had shared their emotions with friends and family members.
  Arms: Supportive Therapy Intervention

SUMMARY:
The present study aims to evaluate whether an online, self-administered, single session intervention (SSI) increases children and adolescents' perceptions of control over external threats and their emotional experience and reduces self-reported symptoms of anxiety and low mood. Children and adolescents, identified by their parents as having difficulties with low mood or anxiety, will be randomised to receive either the growth mindset of personality intervention or an active comparison condition. Whether parental low mood and anxiety has a moderating impact on outcomes will also be investigated.

DETAILED DESCRIPTION:
Despite considerable evidence for the efficacy of psychological interventions for anxiety and depression in children and young people (CYP) (James et al. 2015; Goodyer, 2017) a significant proportion of CYP fail to access such treatments (Children's Commissioner for England 2016). Reasons for this implementation gap are many but include lack of accessibility to Child and Adolescent Mental Health Services (CAMHS) which are operating with long waiting times, high symptom thresholds and constraints in terms of what they are able to offer (Murphy and Fonagy, 2013). In order to reduce the need to access gap, particularly for young people experiencing symptoms of anxiety and depression but whom may not reach service thresholds, there is a need for the development of novel interventions which are cost-effective and can be disseminated at scale (Milat, King, Bauman, & Redman, 2012; Kazdin 2019). Single session interventions (SSI), particularly those which can be completed without therapist guidance, offer a scalable solution and have been found to be effective for a range of psychological difficulties in CYP (Schleider & Weisz 2017). One such SSI targets the implicit beliefs CYP hold about the malleability of their personality (known as their 'mindset') and has been found to reduce adolescent depressive symptoms and parent-reported anxiety over a 9-month period, relative to an active control condition (Schleider and Weisz, 2018). Investigation into trajectories of change found that changes in anxiety and depression were predicted by immediately post intervention changes in perceived primary and secondary control, indicating a potential underlying mechanism. Replication of these findings, along with exploration of predictors of treatment response and diverse opportunities for implementation is required and is the aim of the present study.

This study will test whether an online, self-administered, growth mindset SSI increases perceived primary and secondary control and reduces symptoms of anxiety and depression in children and adolescents aged between 8 and 16, relative to an active "supportive therapy control" condition. Outcome measures will be completed immediately post intervention. A secondary aim for the study will be to investigate the role of parental symptoms of anxiety or low mood as a potential moderator of treatment outcome. In order to achieve these aims, CYP and their parents or caregivers will be recruited through online advertisements, charities and schools.

ELIGIBILITY:
Inclusion Criteria:

* Young person aged between the ages of 8 and 16 years-old
* Young person has difficulties with low mood or anxiety as identified by a parent or caregiver
* Young person has a parent or caregiver willing to take part in the research
* Both the young person and parent must be able to read and understand English to a level enabling them to access the assessment and intervention

Exclusion Criteria:

- None

Ages: 8 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 150 (Estimated)
Dates: Start 2020-11-10 (Actual); Primary Completion 2022-12-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in Perceived Primary Control Scale for Children; Youth-Report | Immediately pre and post intervention
  The Perceived Primary Control Scale for Children (Weisz, Southam-Gerow, & McCarty, 2001; Weisz, Weiss, Wasserman, & Rintoul, 1987) measures young people's perceived ability to exert control over situations or events by exerting personal effort. The measure includes 24 statements relating to primary control (e.g. "I can make friends with other kids if I really try" or "I cannot get good grades no matter how hard I try") and respondents are required to rate their agreement with the statement on a Likert scale with responses ranging from "very false" to "very true".
Change in Perceived Secondary Control Scale for Children; Youth-Report | Immediately pre and post intervention
  The Perceived Secondary Control Scale for Children (Weisz, Francis, & Bearman, 2010) measures young people's perceived ability to control the psychological impact of situations or events through the use of cognitive and behavioural strategies. Participants are required to rate their degree of agreement (on the same scale as the PCSC) to 20 statements regarding secondary control (e.g. "When something bad happens, I can find a way to think about it that makes me feel better" or "When something bad happens, I keep worrying about how bad it is").

SECONDARY OUTCOMES:
Change in Implicit Theories of Personality Questionnaire; Youth-Report | Immediately pre and post intervention
  Young people are asked to rate the extent to which they agree or disagree with three statements about the malleability of their personality on a scale from 1 (really disagree) to 6 (really agree).
Change in Pediatric Quality of Life Inventory (PEDS-QL) Present Functioning Visual Analogue Scales | Immediately pre and post intervention
  The PEDS QL Present Functioning Visual Analogue Scales (Sherman et al. 2006) include four questions assessing young people's current experience of anxiety, sadness, anger and worry. Young people are provided with a scale with a happy face at one end and a sad face at the other end and are asked to move the slider on the scale to the point which best represents how they are feeling at that moment in time.

OTHER OUTCOMES:
Revised Children's Anxiety and Depression Scale (RCADS); Parent-Report | Completed by parents pre-intervention
  The RCADS is a 47-item questionnaire used to screen for symptoms of depression and anxiety in children and adolescents aged 8-18. The measure yields a Total Anxiety Scale (sum of the 5 anxiety sub scales) and a Total Internalising Scale (sum of all 6 subscales). A t-score is calculated from the raw score with a t-score of 65 meaning that the score is roughly in the top 7% of scores of un-referred young people of the same age (described as borderline clinical) and a t-score of 70 meaning that the score is roughly in the top 2% (described as the clinical threshold.
Patient Health Questionnaire (PHQ-9) | Completed by parents pre-intervention
  The PHQ-9 (Kroenke, Spitzer & Williams, 2001) is a 9-item diagnostic screening tool used to assess for and monitor the presence of depressive symptomatology in adults. The questions, which correspond to the diagnostic criteria in DSM-5, ask respondents to quantify the number of days they have been bothered by certain symptoms over the past two weeks. A higher score indicates greater symptom severity.
Generalized Anxiety Disorders Scale (GAD 7) | Completed by parents pre-intervention
  The GAD-7 (Spitzer et al 2006) is a 7-item questionnaire used to assess for symptoms and severity of generalised anxiety disorder (GAD), however it is also used as a screening tool across anxiety disorders due to the transdiagnostic nature of the items and high degree of comorbidity in anxiety disorders (Kroenke et al 2007). As with the PHQ-9, respondents are asked to rate the frequency of symptoms over the past two weeks. A higher score indicates greater symptom severity.
Participant feedback | Immediately post intervention
  Youth will be asked to complete 4 items about their experience of the intervention (e.g. "I understood the activity") on a 5 point scale ranging from strongly disagree to strongly agree. Participants are also given the opportunity to complete an additional 3 open-ended questions about their experience.

CONTACTS AND LOCATIONS:
Overall Officials: Harriet Clarkson, Principal Investigator — Royal Holloway University
Locations (1):
- Royal Holloway, University of London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Data will be available on reasonable request

REFERENCES:
- [Background] Schleider JL, Weisz JR. Reducing risk for anxiety and depression in adolescents: Effects of a single-session intervention teaching that personality can change. Behav Res Ther. 2016 Dec;87:170-181. doi: 10.1016/j.brat.2016.09.011. Epub 2016 Sep 26. PMID 27697671